CLINICAL TRIAL: NCT00000395
Title: Mechanisms of Antifolate Efficacy in Arthritis
Brief Title: Antifolate Effectiveness in Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: R29AR042674 (NIH); R29AR042674 (NIH); NIAMS-035
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2013-06

CONDITIONS: Rheumatoid Arthritis; Adjuvant Arthritis
Keywords: Rheumatoid arthritis; Lewis rat adjuvant arthritis; Antifolate efficacy; Autoimmunity; Adenosine metabolism; Methotrexate therapy; Skeletal disorder; Dietary supplement; Antiarthritic agent; Folic acid
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Experimental; Autoimmune Diseases | interventions — Methotrexate; Leucovorin; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group 1 - Folinic acid (Experimental): Subjects receiving Methotrexate for 6 weeks and 5 mg of Folinic acid daily for 1 week.
  Interventions: Drug: Methotrexate; Dietary Supplement: Folinic acid
- Group 2: Folic acid (Experimental): Subjects receiving Methotrexate for 6 weeks and 5 mg of Folic acid daily for 1 week.
  Interventions: Drug: Methotrexate; Dietary Supplement: Folic acid

INTERVENTIONS:
Drug: Methotrexate
Dietary Supplement: Folinic acid
  Arms: Group 1 - Folinic acid
Dietary Supplement: Folic acid
  Arms: Group 2: Folic acid

SUMMARY:
This study looks at how the arthritis drug methotrexate works in low doses to treat rheumatoid arthritis. (High doses of methotrexate are used to treat some types of cancer.) Methotrexate blocks the action of the B-vitamin known as folic acid. We are studying the biochemical reactions affected by this vitamin because we think that blocking many of these reactions may be necessary for methotrexate to work in treating rheumatoid arthritis. Through these studies, we hope to gain a better understanding of how this drug and related drugs work as treatments for arthritis.

DETAILED DESCRIPTION:
Low-dose methotrexate therapy suppresses autoimmune arthritis in human and animal models. We hypothesize that the effect of methotrexate in the treatment of rheumatoid arthritis is due to the inhibition of aminoimidazole-carboxamide ribotide transformylase, a folate-dependent enzyme that catalyzes the last step in the de novo biosynthesis of inosine monophosphate. The resulting accumulation of aminoimidazole carboxamide riboside inhibits adenosine deaminase, therefore interfering with normal adenosine metabolism. It is well known that children with adenosine deaminase deficiency have severe combined immunodeficiency syndrome. This suggests that adenosine deaminase activity is key to immune competence and is associated with the mechanism of efficacy in methotrexate therapy of rheumatoid arthritis.

Several studies indicate that supplemental folinic acid (5-formyltetrahydrofolate) used in large doses during low-dose methotrexate therapy for rheumatoid arthritis causes a flare in joint inflammation. However, supplemental folic acid (pteroylglutamic acid) does not lessen the efficacy of the therapy. We further hypothesize that if methotrexate efficacy is driven by aminoimidazole carboxamide ribotide transformylase inhibition, folic acid supplementation should not alter urinary levels of aminoimidazole carboxamide, adenosine, and deoxyadenosine, while folinic acid supplementation should prevent the accumulation of these compounds.

We will test our hypotheses both in people with rheumatoid arthritis and in Lewis rat adjuvant arthritis. Our objectives include: (1) determining if the dose level of methotrexate that is clinically optimal in the treatment of Lewis rat adjuvant arthritis interferes with normal adenosine metabolism; (2) determining the effectiveness of drugs that interfere with adenosine metabolism (deoxycoformycin, aminoimidazole carboxamide, and aminoimidazole carboxamide with a suboptimal dose of methotrexate) in Lewis rat adjuvant arthritis; and (3) determining whether supplemental folic acid and folinic acid during methotrexate therapy normalize adenosine metabolism in patients with rheumatoid arthritis. The information we obtain will enhance the understanding of the biochemical action of antifolates/antimetabolites that are effective in the treatment of human and animal arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals starting methotrexate for rheumatoid arthritis.
* Study subjects should not currently be taking folic acid-containing vitamins.

Exclusion Criteria:

* Cancer, renal, or liver disease.
* Previous use of methotrexate within the past 6 months or current use of folic acid-containing supplements.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1996-09; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Determine the effect of Folic acid and Folinic acid on urinary 5-amino=imidazole-4-carboxaminde (AICA in individuals with rheumatoid arthritis treated with low dose methotrexate.

SECONDARY OUTCOMES:
Determine the effect of folic acid and folinic acid on urinary adenosine excretion in individuals with rheumatoid arthritis treated with low dose methotrexate
Correlate disease activity with urinary AICA and adenosine levels

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L. Morgan, M.D., R.D., Principal Investigator — University of Alabama Department of Nutrition Sciences
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Morgan SL, Baggott JE, Vaughn WH, Young PK, Austin JV, Krumdieck CL, Alarcon GS. The effect of folic acid supplementation on the toxicity of low-dose methotrexate in patients with rheumatoid arthritis. Arthritis Rheum. 1990 Jan;33(1):9-18. doi: 10.1002/art.1780330102. PMID 2405864
- [Background] Morgan SL, Baggott JE, Refsum H, Ueland PM. Homocysteine levels in patients with rheumatoid arthritis treated with low-dose methotrexate. Clin Pharmacol Ther. 1991 Nov;50(5 Pt 1):547-56. doi: 10.1038/clpt.1991.180. PMID 1934868
- [Background] Morgan SL, Hine RJ, Vaughn WH, Brown A. Dietary intake and circulating vitamin levels of rheumatoid arthritis patients treated with methotrexate. Arthritis Care Res. 1993 Mar;6(1):4-10. doi: 10.1002/art.1790060103. PMID 8443257
- [Background] Morgan SL, Baggott JE, Vaughn WH, Austin JS, Veitch TA, Lee JY, Koopman WJ, Krumdieck CL, Alarcon GS. Supplementation with folic acid during methotrexate therapy for rheumatoid arthritis. A double-blind, placebo-controlled trial. Ann Intern Med. 1994 Dec 1;121(11):833-41. doi: 10.7326/0003-4819-121-11-199412010-00002. PMID 7978695
- [Background] Morgan SL, Anderson AM, Hood SM, Matthews PA, Lee JY, Alarcon GS. Nutrient intake patterns, body mass index, and vitamin levels in patients with rheumatoid arthritis. Arthritis Care Res. 1997 Feb;10(1):9-17. doi: 10.1002/art.1790100103. PMID 9313385
- [Background] Morgan SL, Baggott JE, Alarcon GS. Methotrexate in rheumatoid arthritis: folate supplementation should always be given. BioDrugs. 1997 Sep;8(3):164-75. doi: 10.2165/00063030-199708030-00002. PMID 18020507
- [Background] Morgan SL, Baggott JE, Lee JY, Alarcon GS. Folic acid supplementation prevents deficient blood folate levels and hyperhomocysteinemia during longterm, low dose methotrexate therapy for rheumatoid arthritis: implications for cardiovascular disease prevention. J Rheumatol. 1998 Mar;25(3):441-6. PMID 9517760
- [Background] Baggott JE, Morgan SL, Koopman WJ. The effect of methotrexate and 7-hydroxymethotrexate on rat adjuvant arthritis and on urinary aminoimidazole carboxamide excretion. Arthritis Rheum. 1998 Aug;41(8):1407-10. doi: 10.1002/1529-0131(199808)41:83.0.CO;2-H. PMID 9704638
- [Background] Strand V, Morgan SL, Baggott JE, Alarcon GS. Folic acid supplementation and methotrexate efficacy: comment on articles by Schiff, Emery et al, and others. Arthritis Rheum. 2000 Nov;43(11):2615-6. doi: 10.1002/1529-0131(200011)43:113.0.CO;2-A. No abstract available. PMID 11083294
- [Background] Alarcon GS, Morgan SL. Guidelines for folate supplementation in rheumatoid arthritis patients treated with methotrexate: comment on the guidelines for monitoring drug therapy. Arthritis Rheum. 1997 Feb;40(2):391; author reply 391-2. doi: 10.1002/art.1780400229. No abstract available. PMID 9041955
- [Background] Morgan SL, Alarcon GS, Moreland L. Improved methotrexate patient information. Arthritis Rheum. 1995 Jun;38(6):874-5. doi: 10.1002/art.1780380633. No abstract available. PMID 7779139
- [Background] Morgan Sl, Alarcon GS, Krumdieck CL. Folic acid supplementation during methotrexate therapy: it makes sense. J Rheumatol. 1993 Jun;20(6):929-30. No abstract available. PMID 8350325
- [Result] Morgan SL, Oster RA, Lee JY, Alarcon GS, Baggott JE. The effect of folic acid and folinic acid supplements on purine metabolism in methotrexate-treated rheumatoid arthritis. Arthritis Rheum. 2004 Oct;50(10):3104-11. doi: 10.1002/art.20516. PMID 15476202